CLINICAL TRIAL: NCT06004076
Title: Effect of Release of Upper Track of Deep Front Fascial Line on Upper Cross Syndrome.
Brief Title: Fascial Release on Upper Cross Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Hussein Mostafa Mahmoud, physiotherapy practitioner, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCS
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Release of upper track of deep front fascial line and supervised corrective exercises
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Release Group (Experimental): Release of upper track of deep front fascial line
  Interventions: Other: Release of upper track of deep front fascial line; Other: Corrective exercises for upper crossed syndrome
- Corrective Group (Other): Corrective exercises for upper crossed syndrome.
  Interventions: Other: Corrective exercises for upper crossed syndrome

INTERVENTIONS:
Other: Release of upper track of deep front fascial line — I will work on upper track of deep front fascial line, I will make release to diaphragm,mediastinum,scalene muscles, scalene fascia,Fascia endothoracic, transversus thoracis,Infrahyoid muscles, fascia pretracheal and Suprahyoid muscles.
  Arms: Release Group
Other: Corrective exercises for upper crossed syndrome — strength for scapular muscles and deep neck flexor

SUMMARY:
This study will be a randomized controlled trial conducted to investigate the effect of release of upper track of deep front fascial line on patients with Upper Cross Syndrome.A sample size of 40 will be randomly allocated to two group ,(20 participants in each group), by using computer-generated random number list method.

Experimental group will receive release of upper track of deep front fascial line in addition supervised corrective exercises for upper crossed syndrome and Control group which will receive supervised corrective exercise only. Both groups will receive eight sessions (2 sessions per week for 4 weeks).

DETAILED DESCRIPTION:
Upper Cross Syndrome is a characterized by muscular imbalance of skeletal muscles activation and inhibition rather than just single muscle involvement. Individuals who present with upper crossed syndrome will show a forward head and neck posture Working in abnormal posture for prolonged duration is the main risk factor.

Although this posture does not necessarily lead to pain, but when prolonged, individuals do often experience upper back and neck pain.Stress on cervico-cranial and Cervico-thoracic junction is caused by the poor posture .Some postural patterning of forward shoulders, increases kyphosis, forward head posture, and loss of cervical lordosis is created by this poor posture.

Many researches studied effect of Exercises, stretching ,muscle energy technique,active release technique.Research on fascia gains more and more attention in basic science.

Fascial tissue plays an important role not only in functional anatomy,but also in sport and exercise science as well as in numerous therapeutic approaches as well as in clinical rehabilitation.Accordingly,There is no studies in the literature investigated the the effect of release of upper anterior track of deep front fascial line in subjects with upper cross syndrome, therefore this is the purpose study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 40 years.
2. Body Mass Index ≤30 kg/m².
3. All participants have forward head ,craniovertebral angle less than 48-50 degrees.
4. All participants have round back(kyphosis angle ≥ 42°).
5. The subjects were chosen from both genders.
6. Based on assessment for upper cross syndrome by photogrammetric analysis

Exclusion Criteria:

1. History of trauma or surgery in cervical region.
2. Bone fractures or acute soft tissue injuries .
3. Osteoporosis .
4. Heart attack .
5. Unstable angina pectoris .
6. Implanted pacemaker or defibrillator .
7. Pregnant women.
8. Cancer .
9. Rheumatoid arthritis.
10. Connective tissue disease: This includes diseases such as osteomyelitis, lupus and scleroderma.
11. Neurological conditions.

    -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Neck disability index | up to 4 weeks
  The neck disability index (NDI) is the most widely used and validated instrument to assess the impact of neck pain on the patient's functional activities and to measure outcomes in clinical practice and research.
  Each of the 10 items scores from 0 to 5. The maximum score is 50. The obtained score can be multiplied by two to produce a percentage score.
  The disability categories for NDI are 0-8%, no disability; 10-28%, mild; 30-48%, moderate; 50-64%, severe; and 70-100%, complete dysfunction.
Craniovertebral angle (CVA) | up to 4 weeks
  The CVA is the angle between a horizontal line passing through the spinous process of C7, and a line extending from the tragus of the ear to C7.
  Photogrammetric analysis will be used to measure the angle.A lateral photograph of the craniocervical region were taken simultaneously from each subject's lateral side view,the distance between the camera and subject will be 150 cm, and the height of the camera will be held at the shoulder height of each subject and each subject will be told to stand in their bare feet.
  The subjects were instructed to fix their eyes on a marker that was attached to the front wall at height of eye while they were comfortably standing straight. were then instructed to assume their natural standing position on a paper sheet barefoot .
  Then, using the USC software application, the angle of the line connecting the tragus and the seventh neck vertebra with the perpendicular line is the forward head angle.

SECONDARY OUTCOMES:
Thoracic kyphosis angle | up to 4 weeks
  To measure the angle of the kyphosis from the bone marker of the spinous process of the seventh vertebra will be used as the starting point of the arc and the spinous process of the 12th dorsal vertebra, T12, was used as the endpoint of the arch .Then, three photos are taken in three numbers using the camera. Then, the digital photos are transferred to the computer and are analyzed using the USC software application.
  Finally, the mean of three measurements is considered as the alignment angle.This method has a high correlation coefficient with the Cobb angle (0.83, 0.89) and precise.
Chest expansion | up to 4 weeks
  The tape-measure will be used for measuring thoracic expansion. Chest expansion, defined as the difference in thoracic girth after maximum inspiration and maximum expiration, is one indicator of chest wall mobility.
  The upper Chest expansion measurements is more useful in clinical practice to evaluate chest mobility and to give indirect information on lung volume function and inspiratory muscle strength.The anatomical marks for upper thoracic expansion are the third intercostal space, the middle of the clavicular line, and spinous process of the fifth thoracic vertebrae.
  The anatomical marks for lower thoracic expansion are the xiphoid process and spinous process of the 10th thoracic vertebrae.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt